CLINICAL TRIAL: NCT02010151
Title: Population Based Intervention Trial of Dispatcher-Activated Neighborhood Access Defibrillation and Cardiopulmonary Resuscitation
Brief Title: Dispatcher-Activated Neighborhood Access Defibrillation and Cardiopulmonary Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korean Center for Disease Control and Prevention (Other Government); Seoul Metropolitan Government Health and Welfare Office (Unknown); Seoul Metropolitan Fire and Disaster Headquater (Unknown); Korea Association for Safety Community (Unknown)
Responsible Party: Principal Investigator, Sang Do Shin, Associated Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SNUEMS201309
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Out of Hospital Cardiac Arrest
Keywords: Out of Hospital Cardiac Arrest; Cardiopulmonary Resuscitation; dispatch; emergency medicine
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAD-CPR (Experimental): When dispatcher detects a patient with OHCA, the dispatcher activates trained neighborhoods by informing events nearby using short message service via cellular phone. The neighborhood within geographically accessible area who could perform effective CPR and defibrillation would be alerted with event of OHCA and the nearest AED.
  Interventions: Other: NAD-CPR
- Conventional dispatcher assisted CPR (No Intervention): When dispatcher detects OHCA, they instruct the caller with CPR instructions. This is conventional dispatcher assisted CPR performed in Seoul.

INTERVENTIONS:
Other: NAD-CPR — When Dispatcher detects OHCA, short message service (SMS)about the OHCA event and information about the location of nearest AED is sent to trained laypersons within geographically accessible area.
  Arms: NAD-CPR

SUMMARY:
The hypothesis of this study is Dispatcher-Activated Neighborhood Access Defibrillation and Cardiopulmonary Resuscitation (NAD-CPR) would improve survival of out-of-hospital cardiac arrest (OHCA).

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) is a major health problem, occurring in about 1 in 1,500 adults in the developed countries each year. Although layperson CPR and defibrillation are crucial components of chain of survival, layperson CPR rate and it's quality is low and public-access defibrillation (PAD) program is not cost-effective.If trained bystanders can know the information of occurrence of OHCA and nearest place for automated external defibrillator (AED) at the same time by dispatch center, these neighborhoods could run and give high quality CPR and early defibrillation. If this protocol ,Dispatcher-Activated Neighborhood Access Defibrillation and Cardiopulmonary Resuscitation(NAD-CPR), is introduced to community, it may improve survival of OHCA.

ELIGIBILITY:
Inclusion Criteria:

* all OHCA with presumed cardiac etiology more than 15 years old
* assessed by emergency medical service (EMS) providers dispatched by dispatch center
* dispatcher detected OHCA patients

Exclusion Criteria:

* OHCA with non-cardiac etiology
* prolonged cardiac arrest with a suspected duration more than 30 minutes
* cases with rigor mortis or rivor mortis, decapitated or decomposed body
* Non detected cases by dispatcher

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3194 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Do Shin, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul Metropolitan City, Seoul, South Korea

REFERENCES:
- [Derived] Lee SY, Shin SD, Lee YJ, Song KJ, Hong KJ, Ro YS, Lee EJ, Kong SY. Text message alert system and resuscitation outcomes after out-of-hospital cardiac arrest: A before-and-after population-based study. Resuscitation. 2019 May;138:198-207. doi: 10.1016/j.resuscitation.2019.01.045. Epub 2019 Mar 19. PMID 30902689

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Dispatcher Assisted CPR: patients enrolled in period that conventional dispatcher assisted CPR was provided to patient (January 2013 to April 2015).
  baseline EMS assessed OHCA: 2,418
  * Adult
  * presumed cardiac etiology
  * Resuscitation attempted
  * Not witnessed by EMS provider
  * Eligible for analysis Final population : 1498
- NAD-CPR: patients enrolled in period that NAD-CPR was provided to patient (May 2015 to December 2017)
  baseline EMS assessed OHCA: 2,611
  * Adult
  * presumed cardiac etiology
  * Resuscitation attempted
  * Not witnessed by EMS provider
  * Eligible for analysis Final population : 1,696 (TM sent: 598)
Period: Overall Study
Arm/Group | Conventional Dispatcher Assisted CPR | NAD-CPR
Started | 1498 (January 2013 to December 2017) | 1696 (January 2013 to December 2017)
Completed | 1498 (Text message (TM) sent: 0) | 1696 (TM sent: 598)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: in the before/after intervention period (January 2013 to April 2015, May 2015 to December 2017), Those cases without an attempted resuscitation effort, cases that were witnessed by EMS providers or those that occurred at a nursing home or medical facility were excluded.
  * both arm participants are not double counted.
Groups:
- Conventional Dispatcher CPR: patients enrolled in period that conventional dispatcher CPR was provided to the patients.
- NAD-CPR: patients enrolled in period that NAD-CPR was provided to the patients.
- Total: Total of all reporting groups
Arm/Group | Conventional Dispatcher CPR | NAD-CPR | Total
Number analyzed (Participants) | 1498 | 1696 | 3194
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [58 to 80] | 72 [59 to 80] | 72 [58 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 532 | 577 | 1109
  Male | 966 | 1119 | 2085
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 1498 | 1696 | 3194
TM sent [Count of Participants; unit: Participants] — TM means text message sent to the volunteers. In Seoul, dispatcher asked two key questions regarding altered mental status and abnormal breathing for suspected arrest according to the DA-CPR protocol. When a cardiac arrest was suspected, the dispatchers pushed a button to send a short text message containing the location of the arrest and nearest PAD to registered volunteers within the same geographic neighborhood.
  Participants | 0 | 598 | 598

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Surviving at Hospital Discharge
Description: we compared the survival to discharge rate between before intervention period and intervention period.
  Survival to discharge checked at the discharge point of hospital.
Time Frame: discharge time from first admission from emergency department within 2 month
Population: Study population excluding exclusion criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Dispatcher CPR | NAD-CPR
Number analyzed (Participants) | 1498 | 1696
Participants | 135 | 216

2. Secondary Outcome: Number of Participants With Pre-Hospital Return of Spontaneous Circulation (ROSC)
Description: we compared the Pre-hospital return of spontaneous circulation (ROSC) rate between before intervention period and intervention period.
Time Frame: hospital arriving time from ambulance within 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Dispatcher CPR | NAD-CPR
Number analyzed (Participants) | 1498 | 1696
Participants | 107 | 223

3. Secondary Outcome: Number of Participants With Good Neurological Recovery
Description: Cerebral performance category 1 or 2 is defined as good neurological recovery. we compared the good neurological recovery rate between before intervention period and intervention period.
Time Frame: discharge time from first admission from emergency department within 2 month
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Dispatcher CPR | NAD-CPR
Number analyzed (Participants) | 1498 | 1696
Participants | 68 | 140

ADVERSE EVENTS:
Time Frame: from hospital arrival (from ambulance) to the hospital or ED discharge within 2 month (All patients have different time frame because all patients have different admission period)
Arm/Group | Conventional Dispatcher CPR | NAD-CPR
All-Cause Mortality (participants affected / at risk) | 1363/1498 | 1480/1696
Serious Adverse Events (participants affected / at risk) | 1363/1498 | 1480/1696
Other Adverse Events (participants affected / at risk) | 0/1498 | 0/1696
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Dispatcher CPR (N=1498) | NAD-CPR (N=1696)
death (Cardiac disorders) | 1363 (1363) | 1480 (1480) — death

LIMITATIONS AND CAVEATS:
It's not randomized trial, it's before-after study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/51/NCT02010151/Prot_SAP_000.pdf